CLINICAL TRIAL: NCT04689425
Title: The Efficacy and Safety of Umbilical Cord Blood Mononuclear Cell Gel in the Treatment of Refractory Diabetic Foot Ulcer.
Brief Title: Umbilical Cord Blood Mononuclear Cell Gel in the Treatment of Refractory Diabetic Foot Ulcer
Acronym: DFU-MNC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Long Zhang, Chief Surgeon, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Long2020-DFU-MNC
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Umbilical cord blood mononuclear cells
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MNC+PRP (Experimental): The combination of PRP and MNC
  Interventions: Drug: Umbilical cord blood mononuclear cell gel（MNC）; Drug: The platelet rich plasma（PRP）
- PRP (Active Comparator): PRP alone.
  Interventions: Drug: The platelet rich plasma（PRP）

INTERVENTIONS:
Drug: Umbilical cord blood mononuclear cell gel（MNC） — Local wound treatment by combination of PRP and MNC, once;
  Other Names: MNC+PRP
  Arms: MNC+PRP
Drug: The platelet rich plasma（PRP） — Local wound treatment by PRP alone, once.
  Other Names: PRP

SUMMARY:
Umbilical cord blood mononuclear cells (MNC) may improve the wound repair ability. This study aims to investigate the role of MNC in refractory diabetic foot ulcer by comparing the combination of PRP and MNC with PRP alone.

DETAILED DESCRIPTION:
The difficulty in the healing of diabetic foot is related to the loss of local repair microenvironment. The platelet rich plasma (PRP) can improve the repair ability, however, the requirement for wound bed preparation is strict, or treatment failure may occur. Umbilical cord blood mononuclear cells (MNC) may provide a better repair environment through paracrine action. This study aims to investigate the role of MNC in refractory diabetic foot ulcer by comparing the combination of PRP and MNC with PRP alone.

ELIGIBILITY:
Inclusion Criteria:

1. The age of the patients is 18-80 years old;
2. Diabetic foot is diagnosed and Wagner grade is above Ⅱ;
3. The duration of ulcer is 2 months or more, with no healing trend for 2 weeks or more.
4. Fasting blood glucose ≤ 9mmol / L, 2 hours postprandial blood glucose ≤ 13mmol / L;
5. The skin oxygen partial pressure around the wound is more than 20mmHg;
6. Sign written informed consent.

Exclusion Criteria:

1. Acute spreading infection of the wound, e.g. massive exudation, redness, swelling, heat, pain.
2. Acute myocardial infarction, heart failure, hepatitis;
3. Active bleeding or hematoma in the wound;
4. Serum albumin <25g/L;
5. Hemoglobin <80g/L;
6. Platelets <50×109/L;
7. Poor cooperate or compliance;The patient cannot cooperate or is.
8. Mentally disabled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound area reduction rate | one week
  The ratio of the reduced area after one week of treatment to the original area

SECONDARY OUTCOMES:
Wound healing rate at 4 weeks | 4 weeks
  Percentage of patients with healed wound at 4 weeks
Amputation rate at 8 weeks | 8 weeks
  Percentage of patients with major amputation at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Long Zhang, Dr., Principal Investigator — Peking University Third Hospital Wound Healing Center
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication, for 1 year
Access Criteria: The IPD and supporting information will be shared by contact PI (Long Zhang)'s Email, upon the request of the scientific journal editor.